CLINICAL TRIAL: NCT06046820
Title: The ENERGY 3 Study: A Randomized, Controlled, Open-Label, Phase 3 Study to Evaluate the Efficacy and Safety of INZ-701 in Children With Ectonucleotide Pyrophosphatase/Phosphodiesterase 1 (ENPP1) Deficiency
Brief Title: The ENERGY 3 Study: Evaluation of Efficacy and Safety of INZ-701 in Children With ENPP1 Deficiency
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Inozyme Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INZ701-106
Record Dates: First submitted 2023-08-28; First posted 2023-09-21 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Ectonucleotide Pyrophosphatase/Phosphodiesterase1 Deficiency; Autosomal Recessive Hypophosphatemic Rickets; Generalized Arterial Calcification of Infancy
Keywords: Ectonucleotide Pyrophosphatase/Phosphodiesterase1 Deficiency; Hypopyrophosphatemia; ENPP1; Autosomal Recessive Hypophosphatemic Rickets Type 2; ARHR2; Generalized Arterial Calcification of Infancy; GACI
MeSH Terms: conditions — Hypophosphatemic Rickets, Autosomal Recessive, 1; Arterial calcification of infancy

STUDY DESIGN:
Intervention Model Description: Study INZ701-106 (ENERGY 3) is a multicenter, randomized in a 2:1 ratio, controlled, open-label Phase 3 study to evaluate the efficacy and safety of INZ-701 in children with ENPP1 Deficiency.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- INZ-701 (Experimental): Subjects randomized to the INZ-701 arm will be administered a 2.4 mg/kg once weekly dose by subcutaneous (SC) injection for the duration of the 52-week Randomized Treatment Period and the Open-label Extension Period.
  Interventions: Drug: INZ-701
- Control Arm (Conventional Therapy) (Active Comparator): Subjects randomized to the control arm will continue taking their conventional therapy as clinically indicated by their treating physician for the duration of the 52-week Randomized Treatment Period.
  Interventions: Drug: Control Arm (Conventional Therapy)

INTERVENTIONS:
Drug: INZ-701 — Recombinant fusion protein that contains the extracellular domains of human ENPP1 coupled with an Fc fragment from an immunoglobulin gamma-1 (IgG1) antibody.
  Other Names: (rhENPP1-Fc).
  Arms: INZ-701
Drug: Control Arm (Conventional Therapy) — Conventional therapy is defined as oral phosphate supplements and calcitriol or other active forms of vitamin D3 (or analogs). No other agents for treatment of ENPP1 Deficiency are allowed in the control arm.
  Arms: Control Arm (Conventional Therapy)

SUMMARY:
The primary purpose of Study INZ701-106 (The ENERGY 3 Study) is to assess the efficacy and safety of INZ-701 in children with ENPP1 Deficiency.

DETAILED DESCRIPTION:
INZ-701 is an ectonucleotide pyrophosphatase/phosphodiesterase 1 (ENPP1) enzyme replacement therapy (ERT) in development for the treatment of ENPP1 Deficiency, an ultra-rare genetic disorder with an incidence of 1 in 64,000 pregnancies.

Study INZ701-106 (The ENERGY 3 Study) is a multi-center, randomized in a 2:1 ratio, controlled, open-label Phase 3 study to evaluate the efficacy and safety of INZ-701 in children with ENPP1 Deficiency.

The study will consist of a Screening Period of up to 52 days (including a washout period of up to 7 days for prohibited medications post-Randomization) and a Randomized Treatment Period (INZ-701 or control) of 52 weeks, followed by an Open-label Extension Period during which all study participants may receive INZ-701, and an End of Study (EOS) Safety visit 30 days after the last dose of INZ-701.

ELIGIBILITY:
Inclusion Criteria

Study participants must meet all of the following inclusion criteria:

1. Caregiver's written or electronic informed consent after the nature of the study has been explained, and prior to any research-related procedures, per International Conference on Harmonisation (ICH) Good Clinical Practice (GCP)
2. Study participant's assent in accordance with local regulations
3. A confirmed postnatal molecular genetic diagnosis of ENPP1 Deficiency with biallelic mutations (ie, homozygous or compound heterozygous) performed by a College of American Pathologists/Clinical Laboratory Improvement Amendments (CAP/CLIA) certified laboratory or regional equivalent
4. Males and females ≥1 year and <13 years of age at Study Day 1
5. Open growth plates of the distal femur and proximal tibia in both legs
6. Plasma PPi concentration of <1400 nM at Screening
7. 25-hydroxyvitamin D (25[OH]D) levels of ≥12 ng/mL at Screening
8. Radiographic evidence of skeletal abnormalities based on an RSS ≥2
9. Female participants of childbearing potential must have a negative serum pregnancy test at Screening and must not be breastfeeding
10. Study participants of childbearing potential who are sexually active must agree to use a highly effective form of contraception in accordance with Clinical Trials Facilitation and Coordination Group (CTFG) guidance and local guidelines for the duration of the study
11. In the opinion of the Investigator, able to complete all aspects of the study

Exclusion Criteria

Study participants meeting any of the following exclusion criteria will not be eligible to participate in the study:

1. In the opinion of the Investigator, has clinically significant disease or laboratory abnormality not associated with ENPP1 Deficiency that will preclude study participation and/or may confound the interpretation of study results
2. If receiving any of the following prohibited medications as indicated in the protocol: systemic corticosteroids (>5 mg prednisone equivalent per day), anti-fibroblast growth factor 23 (FGF23), and oral and/or IV bisphosphonates
3. Unable or unwilling to discontinue calcitriol or other active forms of vitamin D3 (or analogs) within 7 days prior to Study Day 1 and/or oral phosphate supplements within 36 hours prior to Study Day 1 if randomized to the INZ-701 arm
4. Planned orthopedic surgery that may confound the interpretation of study results during the 52-week Randomized Treatment Period
5. Known intolerance to INZ-701 or any of its excipients
6. A positive COVID-19 test within 5 days prior to Randomization, only if required as per local regulations or institutional policy
7. Previous treatment with INZ-701
8. Concurrent participation in another interventional clinical study and/or has received an investigational drug within 5 half-lives of the last dose or within 4 weeks prior to Randomization, whichever is longer, or use of an investigational device

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Plasma Inorganic Pyrophosphate (PPi) concentration through Week 52 | 52 weeks (Baseline through Week 52)
  For each subject, plasma PPi will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.

SECONDARY OUTCOMES:
Change from Baseline in skeletal abnormalities as measured by the Radiographic Global Impression of Change (RGI-C) global score through Week 52 | Baseline, Week 26, Week 52
  The RGI-C is an overall radiographic score which can be used to monitor response to a therapeutic intervention comparing scores from 2 time points. A determination of healing on a scale of 0 to +3 with 0 being no change or healing and +3 being complete healing; worsening is also measured on a scale of 0 to -3 with 0 being no change and -3 being severe worsening.
Change from Baseline in rickets as measured by Rickets Severity Score (RSS) total score through Week 52 | Baseline, Week 26, Week 52
  The RSS assesses rickets severity by utilizing a scoring system that uses a scale from 0 to 4 for the wrists and 0 to 6 for the knees, to generate a total score of 0 to 10, where 0 is normal and 10 is the worst score possible ie, most severe skeletal abnormalities observed radiographically.
Change from Baseline in growth Z-score (height/body length and weight) through Week 52 | Baseline, Day 29, Week 8, Week 13, Week 26, Week 39, Week 52
  A Z-score represents the degree to which that particular measurement for that individual differs from the reference value in the general population.
  (height/body length and weight) through Week 52
Area under the Plasma Concentration versus Time Curve (AUC) of INZ-701 | 52 weeks (Randomized Treatment Period)
  For each subject, variation of concentration of INZ-701 in the plasma will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.
Maximum Plasma Concentration (Cmax) of INZ-701 | 52 weeks (Randomized Treatment Period)
  For each subject, the maximum concentration of INZ-701 in the plasma will be measured via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.
Change from Baseline in ENPP1 activity (µM/min) through week 52 | 52 weeks (Randomized Treatment Period)
  For each subject, the activity of INZ-701 (µM/min) in the serum will be assessed through hydrolysis of a substrate to the enzyme, via a series of blood samples obtained throughout the study, comparing the subject's baseline value over time.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Gunter, MD, Study Director — Inozyme Pharma, Inc.
Locations (15):
- United States (6):
  - Children's Hospital of Colorado, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
- Queensland Children's Hospital, South Brisbane, Australia
- Centre Hospitalier Universitaire (CHU) Sainte-Justine, Montreal, Canada
- Hôpital Bicêtre, Service d'endocrinologie et diabète de l'enfant (Childhood Endocrinology and Diabetes Department), Le Kremlin-Bicêtre, France
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia
- Hospital San Joan de Deu, Barcelona, Spain
- Turkey (Türkiye) (2):
  - Umraniye Training and Research Hospital, Istanbul
  - Cukurova Universitesi Tip Fakultesi, Sarıçam
- Al Jalila Children's Specialty Hospital, Dubai, United Arab Emirates
- Royal Manchester Children's Hospital, Manchester, United Kingdom